CLINICAL TRIAL: NCT04608786
Title: A Single-arm, Open-label，Phase Ib Clinical Study of ZKAB001 Combined With Capecitabine in Adjuvant Therapy for Patients With Biliary Tract Cancer After Radical Resection
Brief Title: A Clinical Study of PD-L1 Antibody ZKAB001 Combined With Capecitabine in Resected Biliary Tract Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTL-LEES-2019-01
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined the therapy using Capecitabine and PD-L1 (Experimental): PD-L1 antibody ZKAB001 D1 5mg/kg every three weeks,up to 16 cycles or 1 year of treatment or the patient has tumor recurrence or metastasis Capecitabine 1000mg / m2/time, 2 times/d for 2 weeks, followed by 1 week of stopping ,three weeks is a course of treatment with a total of 8 courses, or the patient has tumor recurrence or metastasis
  Interventions: Drug: ZKAB001 5mg/kg; Drug: Capecitabine

INTERVENTIONS:
Drug: ZKAB001 5mg/kg — ZKAB001 D1 IV 5mg/kg every three weeks,up to 16 cycles or 1 year
  Other Names: PD-L1 monoclonal antibody
Drug: Capecitabine — Capecitabine po 1000mg / m2/time, 2 times/d for 2 weeks, followed by 1 week of stopping ,three weeks is a course of treatment with a total of 8 courses

SUMMARY:
This is a Phase Ib, open-label,single-arm, clinical study, aiming to investigate the safety, tolerability and pharmacokinetics of ZKAB001 (a fully human monoclonal antibody targeting the Programmed Death - Ligand 1 (PD-L1) membrane receptor ) combined with capecitabine as adjuvant chemotherapy for patients with biliary tract cancers after radical resection.After completing 8 courses of combined treatment ,ZKAB001 was continued to be administered separately once 3 weeks for a total of 16 cycles or 1 year.

DETAILED DESCRIPTION:
This study includes two phases,the first phase is the dose exploration, 6 subjects were first included at the initial dose to confirm the dose safety. If the toxicity is not tolerated, the dose of the chemotherapeutic agent will be reduced depending on the toxicity(including hematological toxicity and non-hematological toxicity) for further exploration. If it can be tolerated, the recommended dose is determined and expanded on this dose. the second phase is the dose expansion, 4 subjects will be enrolled to further observe the safety and efficacy. The DLT(Dose limited toxicity) observation period is set as the first course of treatment(3 weeks). The end point is that the patient has been taking the drug for 16 cycles or 1 year, or the patient dies or develops intolerable toxicity or confirmed disease recurrence or distant metastasis or withdrawal of informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. both men and women, age ≥ 18 years old；
2. A histopathological or cytological diagnosis of gallbladder cancer and extrahepatic cholangiocarcinoma after radical resection
3. Postoperative pathological stage is T2-4 or N1 R0/R1 resection；
4. No more than 12 weeks from radical resection；
5. Eastern Cooperative Oncology Group(ECOG) performance status score 0-1;
6. Estimated life expectancy >6 months;
7. Biliary drainage is in good condition, no current infection ;
8. Have not received radiotherapy, chemotherapy, or immunotherapy for the primary tumor;
9. The function of important organs meets the following requirements:

(1) Blood routine test: absolute neutrophil count (ANC) ≥ 1.5×109/L, platelets ≥ 100×109/L, hemoglobin ≥100g/L; (2) Biochemical tests : ALT, AST ≤ 2.5×ULN; ALB≥ 35g/L;total bilirubin ≤3×ULN; serum creatinine ≤ 1.5×ULN, creatinine clearance rate ≥50 mL/min(Crockcroft-Gault formula); 10.Subjects voluntarily joined the study, signed an informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. Local recurrence or distant metastasis (including ascites or malignant pleural effusion);
2. Severe cardiovascular disease, such as New York Heart Association (New York Heart Association, NYHA standard) heart failure above grade 2, unstable angina, unstable arrhythmia, or color photos of the heart suggest LVEF (left ventricular ejection fraction) )<50%;
3. Known allergy or hypersensitivity to monoclonal antibodies or fluorouracil drugs or their analogues;
4. Subjects with known, active or suspicious autoimmune diseases, who are in a stable state and do not require systemic immunosuppressive therapy can be included in the group;
5. Subjects were treated with immunosuppressants or systemic or absorbable topical corticosteroids within 2 weeks before the first study to achieve immunosuppressive purposes (>10mg/day prednisone or equivalent dose) ;
6. Suffered from other active malignancies within 5 years before the first administration of the study drug. Cured localized tumors, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, etc. can be included in the group;
7. Active viral hepatitis (such as hepatitis B, hepatitis C, unless antiviral treatment is given and the HBV or HCV viral load is below the minimum detection limit can be considered for inclusion), HIV positive or a known history of acquired immunodeficiency syndrome ；
8. Any active infection that requires systemic anti-infective treatment occurs within 14 days before the first medication;
9. Have active tuberculosis in the past 1 year, regardless of treatment;
10. Live attenuated vaccines have been used within 28 days before screening;
11. Subjects who have previously received allogeneic bone marrow transplantation or solid organ transplantation;
12. Have received any other experimental drug treatment within 28 days before signing the ICF;
13. People who have difficulty swallowing or have known drug absorption disorders;
14. Women who are pregnant or breastfeeding;
15. Subjects of childbearing age who refuse to use effective contraceptive measures;
16. Situations that other researchers think are not suitable for inclusion. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 21 days after first dose
  Adverse events of level 3 or above related to the study drug occurring within 21 days after the first dose as assessed by CTCAE v5.0.
Recommended phase II dose (RP2D) | 21 days after first dose
  DLT occurs in no more than 1/6 subjects, this dose is defined as RP2D.

SECONDARY OUTCOMES:
AUC(0-t) | 16 periods or 1 year
  Area under curve 0-t
Cmax | 16 periods or 1 year
  Peak concentration
Tmax | 16 periods or 1 year
  Peak time
Disease-free Survival | up to 24 months
  Form date of randominzation until the date of the first tumor recurrence/ometastasis or death of the subject due to any reason
Overall survival (OS) | up to 24 months
  From date of randomization until the date of death from any cause or the date of last follow-up whichever came first
the number of subjects presenting detectable anti drug antibodies (ADAs) | through study completion,an average of 1 year
  To evaluated the number of subjects presenting detectable anti drug antibodies (ADAs)

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital Affiliated to School of Medicine, Shanghai Jiaotong University, Shanghai, China